CLINICAL TRIAL: NCT05256433
Title: Effectiveness of Instrument Assisted Soft Tissue Mobilization (IASTM) And Manual Massage On Thickness, Pain and Foot Function Among Patient With Plantar Fasciitis
Brief Title: Role of Soft Tissue Therapy in Plantar Fasciitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Hafiza Javeria, Hafiza Javeria Mirza, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ziauddin University
Record Dates: First submitted 2022-02-04; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: INSTRUMENT ASSISTED SOFT TISSUE MOBILIZATION
Keywords: Musculoskeletal Pain; Myofascial Release; Plantar Fasciitis
MeSH Terms: conditions — Musculoskeletal Pain; Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM (Experimental)
  Interventions: Other: Group-A
- Transverse friction massage (Active Comparator)
  Interventions: Other: Group-B

INTERVENTIONS:
Other: Group-A — IASTM Certified IASTM practitioner will be performing the technique with emollient lubricant in which brushing and sweeping stroke will be applied for plantar fascia and fanning and sweeping stroke technique for calf muscles for the duration of 10 minutes to eliminate the inflammation. Active calf stretching and passive plantar fascia stretching will be performed for the correction of shortened tissue, and to prevent re-injury. The frequency stretching will be 5 repetitions for each with 10 seconds hold.
  Arms: IASTM
Other: Group-B — Manual massage includes transverse friction massage for plantar fascia, flexor digitorum brevis, and deep massage for calf muscle for the duration of 10 minutes to eliminate the tightness and increase the blood flow. Active calf stretching and passive plantar fascia stretching will be performed for the correction of shortened tissue, and to prevent re-injury.
  Arms: Transverse friction massage

SUMMARY:
Plantar Fasciitis (PF) is a frequently and commonly reported heel pain present in every age with multifactorial etiology. It is the most common reason for constant heel pain in adults affecting both young active and older sedentary individuals. PF is reported approx. 11%-15% of all foot symptoms demanding professional care among adults. Instrument-Assisted Soft Tissue Massage (IASTM) refers to a technique that utilizes instruments to eliminate scar tissues and work with mending measure through development of new extracellular lattice proteins like collagen that may be effective in providing immediate and quick pain relief by covering a larger area. On the other hand, numerous options with conservative measures has been frequently documented in treating plantar fasciitis that may include stretching, massage, orthosis, anti-inflammatory agents and surgery etc. Although, transverse friction massage has been considered to be one of the best treatment option in reducing pain, releasing tight areas and promoting flexibility. Besides, several studies reported the usefulness of potential assessment tools for remote monitoring of patients that can be utilized by clinicians for wider range of purposes. To the best of author's knowledge, limited studies has been conducted till date utilizing the IASTM technique in comparison to conservative treatment options with standardized assessments in treating PF. Therefore, this study aims to investigate the effectiveness of IASTM to assess thickness, pain, and foot function by using ultrasound for the management of plantar fasciitis patients. The findings of this study may be useful to establish an effective treatment protocol to enhance the quality of life of the target population.

ELIGIBILITY:
Inclusion Criteria:

-Pre-diagnosed adults (18-55 years) with plantar fasciitis of both genders.

Exclusion Criteria:

* Pathological bone spurs of the calcaneus
* Burn scars
* Polyneuropathies
* Corticosteroid injections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
NPRS | Baseline
  It is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
NPRS | 4 weeks
  It is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
FAAM | Baseline
  This self-report outcome instrument is available in English, German, French and Persian. The Foot and Ankle Ability Measure is a 29-item questionnaire divided into two subscales: the Foot and Ankle Ability Measure, 21-item Activities of Daily Living Subscale and the Foot and Ankle Ability Measure, 8-item Sports Subscale.
FAAM | 4 weeks
  This self-report outcome instrument is available in English, German, French and Persian. The Foot and Ankle Ability Measure is a 29-item questionnaire divided into two subscales: the Foot and Ankle Ability Measure, 21-item Activities of Daily Living Subscale and the Foot and Ankle Ability Measure, 8-item Sports Subscale.
Diagnostic Ultrasound | Baseline
  Ultrasound imaging is a noninvasive technique, that uses sound waves to produce pictures of muscles, tendons, ligaments, nerves and joints throughout the body. Ultrasound is extensively used in the radiological department now it is being utilized in the diagnosis of Musculoskeletal related conditions and increasingly being used as an extension to physical examination. In plantar fasciitis, it is used for the measurement of plantar fascia.In symptomatic patients measured <4mm mm in comparison with asymptomatic patients 2.3-4 mm with hyperechoic in nature.
Diagnostic Ultrasound | 4 weeks
  Ultrasound imaging is a noninvasive technique, that uses sound waves to produce pictures of muscles, tendons, ligaments, nerves and joints throughout the body. Ultrasound is extensively used in the radiological department now it is being utilized in the diagnosis of Musculoskeletal related conditions and increasingly being used as an extension to physical examination. In plantar fasciitis, it is used for the measurement of plantar fascia.In symptomatic patients measured <4mm mm in comparison with asymptomatic patients 2.3-4 mm with hyperechoic in nature.

CONTACTS AND LOCATIONS:
Locations (1):
- Javeria Mirza, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No